CLINICAL TRIAL: NCT02992756
Title: Influence of PRGF (Plasma Rich in Growth Factors) Puncture in Ovaries With Low Follicular Reserve
Brief Title: Influence of PRGF (Plasma Rich in Growth Factors) Puncture in Ovaries With Low Follicular Reservetechniques
Acronym: PRGFO-2020
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Due to the difficulty in meeting the selection criteria by preventing continued recruitment to the trial. This has made recruitment more difficult and has prolonged the recruitment time to more than two years from the initially planned end of study
Sponsor: IVI Bilbao (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1607-BIO-057-MF
Record Dates: First submitted 2016-12-02; First posted 2016-12-14 (Estimated); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Low Ovarian Reserve
MeSH Terms: interventions — Intercellular Signaling Peptides and Proteins

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Instillation of growth factors (Experimental): Patients candidates to an IVF/ICSI cycle with low follicular reserve: after at least one cycle of stimulation obtaining 0-3 oocytes.
  Interventions: Drug: Growth Factors

INTERVENTIONS:
Drug: Growth Factors — one dose 3-6 mL of PRP obtained by PRGF Endoret

SUMMARY:
Assisted reproduction patients candidates to an IVF/ICSI cycle with low follicular reserve: after at least one cycle of stimulation obtaining 0-4 oocytes.

Improve the follicular response in patients with low response, increasing the number of follicles in subsequent cycles to treatment with growth factors.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must give written consent.
2. To be a healthy woman acting voluntarily, aged 18 to 42 years (both inclusive) at the time of study selection time of selection for the study.
3. Have a BMI ≥ 18 kg/m2 and ≤ 35 kg/m2
4. Patients with low ovarian reserve (AMH <1.1 ng/mL) according to the Bologna criteria.
5. Patients who are going to undergo IVF/ICSI cycle with low follicular response: who after a previous cycle of stimulation have obtained 0-3 or more follicular 0-3 oocytes have been obtained after a previous stimulation cycle; or if 0-3 oocytes are expected to be obtained at the present time (less than 4 follicles).

   oocytes (less than 4 follicles in the basal ultrasound).
6. To have recent analytical results (haemogram, biochemistry and coagulation); at least 11 months prior to inclusion in the study and a serology, according to clinical practice.

Translated with www.DeepL.com/Translator (free version)

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2021-06-29 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Number of follicles recruited after instability of ovarian growth factors | two months; Time included in two protocols of ovarian stimulation
  o demonstrate an increase of at least 20% in the number of MII oocytes in a cycle after IVF/ICSI treatment with PRGF®-Endoret® compared to previous cycles in low IVF/ICSI patients.
  IVF/ICSI treatment with PRGF®-Endoret® with respect to previous cycles in low responders.
  responders

SECONDARY OUTCOMES:
Rates of pregnancy rates | three months after embryo transfer after treatment of growth factors
  Increase pregnancy rates and decrease the number of cycles of accumulation of oocytes.

CONTACTS AND LOCATIONS:
Locations (1):
- IVI Bilbao, Leioa, Vizcaya, Spain

IPD SHARING:
Plan to Share IPD: No